CLINICAL TRIAL: NCT03709927
Title: A Phase 1, Randomized, Blinded, Placebo and Moxifloxacin Controlled, 4-Period Crossover, Study Evaluating the Effect of ZTI-01 on 12-Lead Electrocardiogram Parameters in Healthy Adult Subject
Brief Title: 4-way Crossover QT Evaluation in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nabriva Therapeutics AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: ZTI-01-101
Record Dates: First submitted 2018-05-08; First posted 2018-10-17 (Actual); Last update posted 2019-03-06 (Actual); Status verified 2019-03

CONDITIONS: Cardiac Repolarization in Healthy Subjects
MeSH Terms: interventions — Fosfomycin; Injections; Moxifloxacin

STUDY DESIGN:
Intervention Model Description: 4-way cross over (two doses of ZTI-01, placebo and oral moxifloxacin)
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Single dose study treatments will be administered in blinded, randomized sequence in separate periods with each subject in the study exposed to each of the four treatments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Therapeutic ZTI-01 6 g IV (Experimental): intravenous fosfomycin (only antibiotic in phosphonic acid derivative class) 6g
  Interventions: Drug: ZTI-01
- Supra-therapeutic ZTI-01 12 g IV (Experimental): intravenous fosfomycin (only antibiotic in phosphonic acid derivative class) 12g
  Interventions: Drug: ZTI-01
- moxifloxacin 400 mg PO (Active Comparator): oral moxifloxacin 400mg film coated tablets - Avelox(TM)
  Interventions: Drug: Moxifloxacin 400mg; Other: Placebo IV
- Placebo IV (Placebo Comparator): IV 0.9% normal saline solution
  Interventions: Other: Placebo IV

INTERVENTIONS:
Drug: ZTI-01 — 6g IV fosfomycin
  Other Names: IV fosfomycin; fosfomycin disodium; fosfomycin for injection
  Arms: Supra-therapeutic ZTI-01 12 g IV; Therapeutic ZTI-01 6 g IV
Drug: Moxifloxacin 400mg — oral moxifloxacin (Avelox 400 mg) + IV normal saline (Placebo)
  Other Names: Positive control
  Arms: moxifloxacin 400 mg PO
Other: Placebo IV — IV Placebo (0.9% Normal Saline)
  Other Names: Negative Control
  Arms: Placebo IV; moxifloxacin 400 mg PO

SUMMARY:
The purpose of this study is to evaluate if ZTI-01 (fosfomycin for injection), an investigational drug being developed to treat people with complicated urinary tract and kidney infections, has any effect on the electrical activity of the heart.

DETAILED DESCRIPTION:
This is a single-center, randomized, placebo-controlled, four-period, cross-over study to assess the effect of single-doses of ZTI-01 at therapeutic (T) and supratherapeutic (ST) plasma concentrations on the QTc interval versus placebo (P) and an open-label moxifloxacin (M) control (400 mg PO).

Assessment of safety data will include changes from baseline in vital signs and laboratory parameters, infusion site reactions, adverse events and clinically significant changes from baseline in 12-lead ECG parameters.

ELIGIBILITY:
Inclusion Criteria:

* physically and mentally healthy volunteer
* a man or woman, 18 to 55 years of age
* a woman of childbearing potential using birth control / negative pregnancy test or a woman of non-childbearing potential
* males with female partners of childbearing potential agree to use contraception
* body mass index 19.0 to 32.0 kg/m2; weight of at least 60.0 kg at Screening
* willing to complete the required 4 study periods

Exclusion Criteria:

* History or evidence of cerebrovascular or cardiac disease
* Uncontrolled hypertension
* Electrographically significant abnormalities on ECG
* Clinically significant medical history (PI assessment)
* Clinically relevant lab abnormalities (PI assessment)
* Calculated eGFR < 60.0 mL/min/1.73m2 based on CKD-EPI 2009 equation
* Abnormal liver tests
* Positive serology HIV, HBsAg, or Hep C virus
* Hemoglobin, hematocrit, electrolytes below lower limit of normal
* Received any hepatic or renal clearance altering agents within 30 days
* History of allergy or hypersensitivity to drugs with clinically significant reaction
* Unwilling to refrain from strenuous exercise from 7 days prior to admission until discharge
* Uses any prescription drug / OTC, within 7 days prior to admission, or 14 days prior to Admission if the drug is a potential inducer or inhibitor of cP450, or 5 half-lives (if longer), or subject continued use of a prescription drug / OTC medication (except contraceptives)
* Scheduled to have surgical procedure during study
* Acute illness that has resolved in less than 14 days, or has had a major illness, or hospitalization within 1 month
* Unwilling to abstain from ingestion of caffeine or xanthine-containing products 96 hours prior and throughout study
* Unwilling to abstain from alcohol beginning 72 hours prior and throughout study
* History of high alcohol consumption within 6 months
* History of drug abuse (in the previous 3 years) or positive urine drug screen
* Used tobacco-containing products within 6 months or has a positive cotinine
* Consumed grapefruit and/or grapefruit juice within 14 days and throughout study
* Consumed other fruit juices within 72 hours and throughout study
* Consumed cruciferous vegetables or charbroiled meats within 7 days and throughout study
* Donated plasma or blood within 30 days or has a history of blood donation of > 450 mL within 3 months
* Used any investigational drug within 30 days
* Previously received fosfomycin
* Deemed by the Investigator to be inappropriate for this study
* Participated in another clinical study within 30 days (or 5 half-lives)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2018-01-11 (Actual); Primary Completion 2018-04-12 (Actual); Study Completion 2018-08-21 (Actual)

PRIMARY OUTCOMES:
Effect of ZTI-01 at the therapeutic and supra-therapeutic plasma concentration on cardiac repolarization expressed by QT interval | 24 hour Holter ECG at Baseline (Day -1) & day of dosing (Day 1) in each of 4 periods. 10 replicates per time point at 13 timepoints: pre-dose: 60, 45 and 30 minutes; after the start of infusion: 0.5, 1 (end infusion), 1.25, 1.5, 2, 3, 4, 8, 12, & 24 hrs
  Determine the change-from-baseline QTc (ΔQTc) when compared with placebo, and moxifloxacin (400 mg PO)

SECONDARY OUTCOMES:
Treatment emergent adverse events (TEAEs) | From Day 1 start of dosing up to Day 36-38 (final follow up visit)
  Number and percentage of subjects reporting a TEAE overall and by treatment

OTHER OUTCOMES:
Cmax after a single dose IV administration of ZTI-01 6g and 12g | Cmax at end of 1-hour single dose infusion
  Maximum plasma concentration Cmax (microg/mL) by dose (6g and 12g)

CONTACTS AND LOCATIONS:
Overall Officials: Evelyn J Ellis-Grosse, PhD, Study Chair — Chief Scientific Officer
Locations (1):
- Pharmaron, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
final report, publication